CLINICAL TRIAL: NCT00244998
Title: Phase II Study of Fulvestrant (Faslodex®) in Androgen Independent Prostate Cancer
Brief Title: Fulvestrant in Treating Patients With Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 53805
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fulvestrant — IM

SUMMARY:
RATIONALE: Estrogen may cause the growth of prostate cancer cells. Hormone therapy using fulvestrant may fight prostate cancer by blocking the use of estrogen by the tumor cells.

PURPOSE: This phase II trial is studying how well fulvestrant works in treating patients with advanced prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if the prostate-specific antigen objective response (complete and partial response) rate is > 0.2 in patients with androgen-independent advanced prostate cancer treated with fulvestrant.

Secondary

* Determine the toxicity of this drug in these patients.

OUTLINE: This is an open-label study.

Patients receive fulvestrant intramuscularly on days 0, 14, and 28. Courses repeat once a month in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for survival.

PROJECTED ACCRUAL: A total of 33 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the prostate

  * Advanced disease
* Must have androgen-independent prostate cancer meeting the following criteria:

  * Evidence of rising prostate-specific antigen (PSA) level and absolute value ≥ 5 ng/mL based on 2 measurements taken ≥ 2 weeks apart (measurements must be done after androgen deprivation [orchiectomy or luteinizing hormone-release hormone (LHRH) analogue] and antiandrogen withdrawal)
* Rising PSA required for ≥ 28 days after antiandrogen or progestational therapy for prostate cancer (≥ 42 days after bicalutamide or nilutamide)
* Testosterone < 50 ng/mL (unless surgically castrated)
* Measurable or evaluable disease

  * PSA elevation constitutes evaluable disease

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC > 3,000/mm^3
* Neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8 g/dL (transfusion or epoetin alfa allowed)
* No bleeding diathesis (e.g., disseminated intravascular coagulation or clotting factor deficiency)

Hepatic

* Bilirubin normal

  * Gilbert's disease with bilirubin ≤ 3 times upper limit of normal (ULN) allowed in the absence of other etiology (e.g., hemolysis-reticulocyte count < 5%) and liver function tests normal
* SGOT and/or SGPT ≤ 2 times ULN
* INR < 1.6

Renal

* Creatinine < 2.5 mg/dL

Cardiovascular

* No unstable cardiac disease requiring medication
* No new onset crescendo or rest angina

  * Stable exertional angina allowed

Other

* Fertile patients must use effective barrier contraception during and for 3 months after completion of study treatment
* No other active malignancy within the past 2 years except nonmelanoma skin cancer or superficial bladder cancer
* No history of significant neurologic or psychiatric disorders, including psychotic disorders, dementia, or seizures
* No other serious illness or medical condition
* No active infection
* No known hypersensitivity to active or inactive excipients of fulvestrant (e.g., castor oil or mannitol)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior retinoids, vaccines, and cytokines are not considered cytotoxic and are allowed

Chemotherapy

* No more than 1 prior cytotoxic chemotherapy regimen
* More than 3 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas)
* No concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* Prior glucocorticoids, antiandrogens, progestational agents, estrogens, and LHRH analogues are not considered cytotoxic and are allowed
* At least 4 weeks since prior flutamide (6 weeks for bicalutamide or nilutamide)
* Concurrent megestrol acetate allowed at a stable dose of ≤ 40 mg/day
* Concurrent androgen deprivation using LHRH analogues allowed but must continue during study treatment or orchiectomy is required to maintain castrate levels of testosterone

Radiotherapy

* More than 3 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* See Endocrine therapy

Other

* Recovered from all prior therapy
* Prior cholecalciferol analogues, ketoconazole, aminoglutethimide, peroxisome-proliferation-activated receptor-gamma agonists or antagonists, or PC-SPES are not considered cytotoxic and are allowed
* No prior long-term anticoagulation therapy (antiplatelet therapy allowed)
* More than 4 weeks since prior investigational drugs
* No other concurrent anticancer therapy (e.g., PC-SPES)
* No concurrent bisphosphonates unless receiving a stable dose at study entry
* No concurrent therapy that may alter androgen metabolism or androgen levels
* No concurrent full anticoagulation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-09; Primary Completion 2006-10 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Prostate-specific antigen (PSA) objective response rate (complete response [CR] or partial response [PR]) | Monthly

SECONDARY OUTCOMES:
Toxicity | Every Month

CONTACTS AND LOCATIONS:
Overall Officials: Donald L. Trump, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States